CLINICAL TRIAL: NCT06371144
Title: A Randomized Control Trial on Intravenous Paracetamol Versus Intramuscular Tramadol as Intra Partum Labor Analgesia in Pregnant Women at Alex Ekwueme Federal University Teaching Hospital Abakaliki
Brief Title: A Randomized Control Trial on Intravenous Paracetamol Versus Intramuscular Tramadol as Intra Partum Labor Analgesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Darlington-Peter Chibuzor Ugoji (Other)
Responsible Party: Sponsor-Investigator, Darlington-Peter Chibuzor Ugoji, Dr, Alex Ekwueme Federal University Teaching Hospital
Organization: Alex Ekwueme Federal University Teaching Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NHREC/16/05/22/130
Record Dates: First submitted 2023-10-16; First posted 2024-04-17 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pain
Keywords: Labour analgesia, paracetamol, tramadol
MeSH Terms: conditions — Pain | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: To compare intravenous paracetamol versus intramuscular tramadol as labour analgesia and to evaluate the incidence of side effects on mother and baby of both drugs
Who Masked: Participant
Masking Description: Double blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paracetamol group (Experimental): Receive intravenous paracetamol intrapartum as labour analgesia
  Interventions: Drug: Paracetamol
- Tramadol group (Active Comparator): Receive intramuscular tramadol intrapartum as labour analgesia
  Interventions: Drug: Paracetamol

INTERVENTIONS:
Drug: Paracetamol — Analgestic
  Other Names: Acetaminophen

SUMMARY:
ABSTRACT BACKGROUND: Labor pain is one of the most excruciating pain experienced by women. It affects maternal psychology and the course of labor causing apprehension, anxiety, and stress. Therefore there is a need for a safe and effective analgesic with minimal maternal and fetal side effects like intravenous paracetamol which has been shown to have great analgesic effect in labour with minimal maternal and neonatal side effects.

OBJECTIVE: To compare intravenous paracetamol versus intramuscular tramadol as labour analgesia and to evaluate the incidence of side effects on mother and baby of both drugs.

METHOD: This would be a hospital based randomized controlled trial comparing intravenous paracetamol to intramuscular tramadol as labour analgesia in pregnant women in active phase of labour in the department of obstetrics and gynecology at Alex-Ekwueme Federal University Teaching Hospital and St. Patrick Mile 4 hospital, Abakaliki. A total of 194 pregnant women in active phase of labour will be included in study after fulfilling the inclusion criteria. These women will be divided into 2 groups of 97 each. Group A will receive a 100ml intravenous infusion containing 1000mg of paracetamol single dose over 15min. Group B: will receive intramuscular tramadol hydrochloride 100mg single dose. Pain intensity of women with both drugs will be noted before administration of drug, one hour, two hours and three hours after administration of drug using the visual analog scale. Perinatal outcome will also be recorded.

10 ANALYSIS AND RESULTS: Data will be collated, tabulated and then statistically analyzed using Statistical Package for Social Science (IBM SPSS) software (version 24, Chicago II, USA). Continuous variables will be presented as mean and standard deviation (Mean ± 2SD) or median and range as appropriate, while categorical variables will be presented as frequencies and percentages. Chi-square test( or Fisher's exact test where applicable) will be used for comparison between groups for categorical variables while student t test or Mann-Whitney U test will be used for comparison between groups for continuous variables KEYWORDS Labour analgesia, intravenous paracetamol, intramuscular tramadol, visual analog scale, neonate, side effects.

DETAILED DESCRIPTION:
METHODOLOGY STUDY DESIGN This will be open label randomized controlled study on the comparison of intravenous paracetamol versus intramuscular tramadol as labour analgesia at the Alex Ekwueme Federal University Teaching Hospital, Abakaliki and St Patrick's Mile 4 Hospital, Abakaliki where both the researcher and trial participants are fully aware of which treatment group the participants are in and what treatments are assigned to them. 3.2. STUDY BACKGROUND The study will be done at the Alex Ekwueme Federal University Teaching Hospital, Abakaliki (AE-FUTHA), Ebonyi state. Ebonyi state is one of the 5 south eastern states in Nigeria. It was created in 1996 and is inhabited predominantly by the Igbo tribe. Abakaliki is the state capital. The state has a population of about 3 million people and occupies a land mass of 5932 kilometers square. Majority of the inhabitants engage in subsistent farming, petty trading and civil service as their occupation. Literacy level generally is low while poverty is prevalent among this population. Alex Ekwueme Federal University Teaching Hospital, Abakaliki (AE-FUTHA) was established in December 2011 following the merger between the defunct Federal medical Centre, Abakaliki and then Ebonyi State University Teaching Hospital, Abakaliki. It receives referrals from all parts of the state and neighboring states of Abia, Benue, Cross-River and Enugu. There are 54 obstetric bed spaces including postnatal and antenatal wards. The hospital runs a busy obstetric unit which is composed of five teams that are subdivided into two units, each unit manned by at least three consultants, senior registrars, registrars and house officers. The department of Obstetrics and Gynecology runs antenatal clinics managed by consultants and resident doctors assisted by trained nurses, midwives and other health workers. The antenatal clinic holds from Monday through Friday with about 5000 antenatal registrations per year. Antenatal clients are booked and assigned to consultants according to the units/teams running antenatal clinic that day. Preliminary data showed that the hospital had 984 deliveries in 2021 with approximately 82 deliveries per month. St. Patrick's Mile 4 Hospital, Abakaliki was established in 1948. It is a missionary hospital managed by Reverend Sisters. It is one of the hospitals in which residents from the AE-FUTHA pass through for their labour ward posting and/or rural posting in obstetrics and gynecology. The obstetrics and gynecology department of the hospital is run by two obstetrician- gynecologists with senior registrars and registrars posted from AE-FUTHA as well as medical officers and the nursing staff. The hospital runs antenatal clinic on Mondays to Wednesdays. It had 2100 deliveries in 2021 with approximately 175 per month.

STUDY SITE The study will be conducted in the labour ward suites of AE-FUTHA and St. Patrick Mile 4 Hospital Abakaliki.

STUDY POPULATION Participants in this study will be drawn from the population of booked women admitted in active phase of labour at the Alex Ekwueme Federal University Teaching Hospital, Abakaliki and St Patrick Mile 4 Hospital, Abakaliki who meet the inclusion criteria. The patients will be selected once they come in active labour (cervical dilatation of greater or equal to 4cm). Parturients will be counseled at the antenatal clinic to present once they start having symptoms of labour. They are usually educated about labour analgesia during the antenatal clinic period and they will be further educated about this particular work by the chief researcher and research assistants. Once the parturient presents in labour and a diagnosis of active labour made, those who meet the inclusion criteria and consented will be recruited into the study. The details of the study they were educated about at the antenatal clinic will be further briefly explained to them before informed consent will be obtained. They will also be assured of confidentiality. A detailed history will be obtained and a thorough examination will be carried out on all the patients in labour. They will be assured of optimal care even if they did not consent to participate in the study

STUDY DURATION The study will last for a period of 3 months. This was extrapolated from the finding that AEFUTHA and St Patrick's Mile 4 Hospital had a total of 3084 labour deliveries in 2021. Approximately 257 labour deliveries per month for both hospitals.

INCLUSION CRITERIA

1. Pregnant women carrying live singleton fetuses at 37-42 weeks' gestational age.
2. Pregnant women in active phase of labour; cervical dilatation ≥ 4cm
3. Spontaneous onset of labour.
4. Singleton pregnancy with vertex presentation

EXCLUSION CRITERIA 1. Women with clinical evidence of cephalopelvic disproportion 2. Malpresentation 3. Multiple pregnancy 4. Previously scarred uterus (post myomectomy, post caesarean) 5. Preterm labour 6. Induced labour 7. Antepartum hemorrhage 8. Pregnancy induced hypertension 9. History of known allergy to tramadol and paracetamol or opioids 10. History of medical disorders 11. Fetal distress 12. Intrauterine fetal death 13. Refusal to give consent STUDY PROCEDURE All the eligible women who had spontaneous active phase labour will be randomized. A proforma form will be filled at the time of admission into the labour ward and antenatal records of the patients will be reviewed, history taking and physical examination will be done, and then those who give informed consent on admission will be enrolled into the study. The socio-demographic data (age, marital status, tribe, religion, occupation, and educational status) and obstetric 35 data of the patients (parity, last menstrual period, and estimated date of delivery), will be collated in the proforma.

Each patient will be further educated about the trial drugs and on the visual analogue scale (VAS) system for the assessment of pain at enrollment. The VAS is a continuous scale comprised of a horizontal or vertical line, 10cm (100mm) in length, anchored by 2-word descriptors at each end (no pain at one end and worst pain at the other end).48 It is self-completed by the respondent who is asked to place a line perpendicular to the VAS line at the point that represents their pain intensity. The patient marks on the line the point that she feels represents the perception of her current pain state. Using a ruler, the score is determined by measuring the distance in millimetres on the 10cm line between the "no pain" anchor and the patient's mark, providing a range of score between 0-100. A higher score indicates greater pain intensity. The following cut off points on the pain VAS have been recommended: no pain (0-4mm), mild pain (5-44mm), moderate pain (45-74mm), and severe pain (75-100mm).41 The marked part is then measured from the left end to determine the actual score. The VAS takes less than 1 minute to complete and is therefore not a burden to a respondent. The patients will be made to know that their involvement will be voluntary and that they could withdraw from participating at any point during the study. They will also be made to understand that if they withdraw from the study, their decision would not affect their subsequent care from the labour ward staff.

Eligible women who present to the labour ward will be consecutively recruited into the study until the required sample size is obtained. The parturients would sign a written consent form before participation. As stated, at the time of admission, history will be taken, the antenatal records of the parturients reviewed and clinical examination will be done. The initial VAS scores will be assessed before randomization, time noted and analgesic administered. Intrapartum monitoring will be done with the individualized partograph according to the departmental protocol. In the labour room, randomization and analgesia will be administered.

A research assistant will be chosen to compute the findings of the study. This research assistant chosen to do this will record the patient's serial number and group in a book that will be provided and which will be kept in the labour ward till the end of the data collection. Rescue or repeat analgesia will be given when patients demands, however, this was another analgesia other than the one from the initial pool {e.g., if patient X who was on analgesia A, requires rescue analgesia, she would be given a rescue analgesia from the pool containing analgesia B}. The amount of this rescue analgesia given will help us know how well the initial analgesia worked and the interpretation of the final results of this study. Labour pain will be assessed at intervals following the initial administration of analgesia (1, 2, and 3 hours after).

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women carrying live singleton fetuses at 37-42 weeks' gestational age.
2. Pregnant women in active phase of labour; cervical dilatation ≥ 4cm
3. Spontaneous onset of labour.
4. Singleton pregnancy with vertex presentation

Exclusion Criteria:

1. Women with clinical evidence of cephalopelvic disproportion
2. Malpresentation
3. Multiple pregnancy
4. Previously scarred uterus (post myomectomy, post caesarean)
5. Preterm labour
6. Induced labour
7. Antepartum hemorrhage
8. Pregnancy induced hypertension
9. History of known allergy to tramadol and paracetamol or opioids
10. History of medical disorders
11. Fetal distress
12. Intrauterine fetal death
13. Refusal to give consent

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Gender Based: Yes — women in labour
Enrollment: 194 (Actual)
Dates: Start 2022-06-03 (Actual); Primary Completion 2022-09-10 (Actual); Study Completion 2022-09-10 (Actual)

PRIMARY OUTCOMES:
Mean pain score | 4hours following administration of each agent
  A standardized scale will be used to asses the mean pain score

CONTACTS AND LOCATIONS:
Overall Officials: OGBO DR UZOMA, MBBS, Principal Investigator — Alex Ekwueme Federal University Teaching Hospital
Locations (1):
- AEFUTHA, Abakaliki, Ebonyi State, Nigeria